CLINICAL TRIAL: NCT03128736
Title: A Pilot Study Comparing Clinical Efficacy of One-Week Dual Delayed-Release Dexlansoprazole 60 mg and Esomeprazole 40 mg for Gastroesophageal Reflux Disease Grade A and B
Brief Title: Comparing Clinical Efficacy of One-Week Dual Delayed-Release Dexlansoprazole and Esomeprazole for GERD Grade A and B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-2014-09-02(I)
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole; Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexlansoprazole group (Experimental): dexlansoprazole 60mg
  Interventions: Drug: Dexlansoprazole group
- esomeprazole group (Experimental): esomeprazole 40mg
  Interventions: Drug: Esomeprazole group

INTERVENTIONS:
Drug: Esomeprazole group — Esomeprazole 40mg qd
  Other Names: Nexium
  Arms: esomeprazole group
Drug: Dexlansoprazole group — Dexlansoprazole 60mg qd
  Other Names: Dexilant
  Arms: dexlansoprazole group

SUMMARY:
Rapid onset of proton-pump inhibitors to achieve a fast symptom is an unmet need in treating gastroesophageal reflux disease (GERD) but there was no report on the short-term clinical effects and timing to symptom relief comparing dexlansoprazole 60 mg to esomeprazole 40 mg. This pilot study aims to compare the one-week clinical effects of single doses of the two drugs in treating GERD patients.

DETAILED DESCRIPTION:
A comparative study to different PPIs in pharmacokinetic change showing that after 12-24 hours post dose, mean percentage of time with pH > 4 and average of mean pH were greater for dexlansoprazole than esomeprazole . However, the study did not report the clinical effect after tablets used. There was no report on the short-term clinical effects and timing to symptom relief of gastroesophageal reflux disease (GERD) between dexlansoprazole 60 mg and esomeprazole 40 mg. Therefore, we conducted a randomized controlled, open-label, study to compare the 7-day clinical effects of single doses of dexlansoprazole 60 mg and esomeprazole 40 mg in for GERD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical symptoms of acid regurgitation, heart burn, or feeling of acidity in the stomach, who have Los Angeles Grade A and B erosive esophagitis proven by endoscopy were recruited

Exclusion Criteria:

* taking antisecretory agents, such as PPIs and histamine-2 receptor antagonists within 2 week prior to the endoscopy
* coexistence of peptic ulcer or gastrointestinal malignancies
* pregnancy
* coexistence of serious concomitant illness (for example, decompensated liver cirrhosis and uremia),
* previous gastric surgery
* allergy to dexlansoprazole or esomeprazole
* symptom score of a validated questionnaire (Chinese GERDQ) less than 12

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of complete symptom resolution (CSR) | 1 week after finishing study drug
  Evaluate the complete symptom resolution by questionnaire

SECONDARY OUTCOMES:
Rate of symptom relapse | 12 weeks after finishing study drug
  Symptom relapse is defined as (a) two or more episodes of reflux symptoms per week that impair the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Deng-Chyang Wu, MD, PhD, Principal Investigator — Kaohsiung Medical University; Seng-Kee Chuah, MD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang HH, Wu DC, Hsu PI, Kuo CH, Tai WC, Yang SC, Wu KL, Yao CC, Tsai CE, Liang CM, Wang YK, Wang JW, Huang CF, Chuah SK; Taiwan Acid-Related Disease Study Group. Clinical efficacy of 60-mg dexlansoprazole and 40-mg esomeprazole after 24 weeks for the on-demand treatment of gastroesophageal reflux disease grades A and B: a prospective randomized trial. Drug Des Devel Ther. 2019 Apr 26;13:1347-1356. doi: 10.2147/DDDT.S193559. eCollection 2019. PMID 31118571